CLINICAL TRIAL: NCT00932698
Title: An Open-Label, Dose-Escalation, Phase 1 Study of the Oral Form of Ixazomib (MLN9708), a Second-Generation Proteasome Inhibitor, in Adult Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study of Oral Ixazomib in Adult Participants With Relapsed and/or Refractory (RR) Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16003; U1111-1177-7936 (Registry Identifier: WHO)
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-06

CONDITIONS: Relapsed and Refractory Multiple Myeloma
Keywords: Relapsed multiple myeloma; Refractory multiple myeloma; Ixazomib Proteasome inhibitor
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 (Experimental): Ixazomib 0.24 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 220 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 (Experimental): Ixazomib 0.48 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 270 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 (Experimental): Ixazomib 0.8 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 137 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 (Experimental): Ixazomib 1.2 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 1436 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 (Experimental): Ixazomib 1.68 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 456 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 (Experimental): Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 1621 days).
  Interventions: Drug: Ixazomib
- Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 (Experimental): Ixazomib 2.23 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months (Up to 2434 days).
  Interventions: Drug: Ixazomib
- Relapsed and Refractory Expansion Cohort: Ixazomib 2 mg/m^2 (Experimental): Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months, Participants must also be refractory to their most recent therapy as evidenced by PD while on therapy or within 60 days after their last dose of therapy (Up to 1621 days).
  Interventions: Drug: Ixazomib
- Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 (Experimental): Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months. Participants with relapsed or refractory disease after >=1 prior therapy but have relapsed after previous Velcade exposure and were not treated with any other proteasome inhibitors (Up to 1573 days).
  Interventions: Drug: Ixazomib
- Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 (Experimental): Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months. Participants with relapsed or refractory disease after >=1 prior therapy which must include thalidomide (or lenalidomide) and corticosteroid, but who never received a proteasome inhibitor (Up to 550 days).
  Interventions: Drug: Ixazomib
- Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2 (Experimental): Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months. Participants who previously received carfilzomib and had relapsed or refractory disease (Up to 123 days).
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: MLN9708

SUMMARY:
This study will determine the safety profile, tolerability, and maximum tolerated dose (MTD) and disease response of Ixazomib administered orally in participants with relapsed and/or refractory multiple myeloma.

DETAILED DESCRIPTION:
The drug being tested in this study is ixazomib. Ixazomib is being tested to treat people who have multiple myeloma. This study will look at the safety and efficacy of ixazomib and will enroll approximately 60 participants.

Participants will receive ixazomib by oral capsule twice weekly on Days 1, 4, 8, and 11 of a 21-day cycle. The study will consist of a dose escalation phase to determine the MTD, followed by an expansion phase in which participants will be treated at the MTD.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 8 years.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

* Multiple myeloma diagnosed according to the standard criteria.
* Participants with multiple myeloma who have relapsed following at least 2 lines of therapy.
* Participants must have measurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
* Male participants who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse.
* Voluntary written consent.
* Suitable venous access for study-required blood sampling.

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Peripheral neuropathy greater than or equal to (>=) Grade 2.
* Female participants who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 14 days before the first dose of study drug.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before the first dose of study treatment.
* Life-threatening illness unrelated to cancer.
* Diarrhea > Grade 1, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) categorization.
* Systemic antineoplastic or radiation therapy within 14 days of cytotoxic agents within 21 days before the first dose of study treatment.
* Treatment with any investigational products within 21 days before the first dose of study treatment.
* Treatment with any investigational proteasome inhibitor.
* Systemic treatment with prohibited medication.
* Ongoing therapy with corticosteroids greater than 10mg of prednisone or its equivalent per day. Inhaled and topical steroids are permitted.
* Central nervous system involvement.
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months.
* Corrected QT interval (QTc) > 470 milliseconds on a 12-lead electrocardiogram (ECG) obtained during the screening period.
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption of tolerance of ixazomib including difficulty swallowing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Gupta N, Yang H, Hanley MJ, Zhang S, Liu R, Kumar S, Richardson PG, Skacel T, Venkatakrishnan K. Dose and Schedule Selection of the Oral Proteasome Inhibitor Ixazomib in Relapsed/Refractory Multiple Myeloma: Clinical and Model-Based Analyses. Target Oncol. 2017 Oct;12(5):643-654. doi: 10.1007/s11523-017-0524-3. PMID 28803351
- [Derived] Richardson PG, Baz R, Wang M, Jakubowiak AJ, Laubach JP, Harvey RD, Talpaz M, Berg D, Liu G, Yu J, Gupta N, Di Bacco A, Hui AM, Lonial S. Phase 1 study of twice-weekly ixazomib, an oral proteasome inhibitor, in relapsed/refractory multiple myeloma patients. Blood. 2014 Aug 14;124(7):1038-46. doi: 10.1182/blood-2014-01-548826. Epub 2014 Jun 11. PMID 24920586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 12 October 2009 to 23 May 2017.
Pre-assignment Details: 60 participants with a diagnosis of relapsed and/or refractory (RR) multiple myeloma were enrolled in 1 of 7 ixazomib dose escalation groups (26 participants) and/or 1 of 4 ixazomib dose expansion groups (40 participants). 6 Participants in 2.0 mg/m^2 dose escalation cohort were also included in the expansion group: 5 in RR, 1 in VR arms.
Groups:
- Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2: Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determined the participant would benefit from therapy beyond 12 months, Participants must also be refractory to their most recent therapy as evidenced by PD while on therapy or within 60 days after their last dose of therapy (Up to 1621 days).
Period: Part 1 (Dose Escalation)
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Started | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 (6 participants from 2.0 mg/m^2 dose cohort transitioned to dose expansion cohort: 5 in RR, 1 in VR.) | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 2 | 2 | 2 | 3 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Participant | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2 (Dose Expansion)
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 12 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 12 | 6 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 8 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of ixazomib. A total of 60 participants participated in the study. There were 7 participants in Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 arm group, 6 out of 7 participated in both phases of the study and were counted once in the expansion cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 1 | 4 | 20 | 12 | 6 | 2 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.02) | 61.3 (6.81) | 69.3 (12.10) | 66.0 (7.00) | 64.0 (9.85) | 78 (NA) — Standard deviation is not estimable for 1 participant. | 64.3 (7.50) | 64.4 (9.58) | 65.4 (8.02) | 64.0 (6.84) | 71.5 (3.54) | 65.2 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 12 | 6 | 1 | 2 | 28
  Male | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 8 | 6 | 5 | 0 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 3 | 2 | 2 | 3 | 3 | 1 | 4 | 20 | 9 | 6 | 2 | 55
  Missing | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 2 | 3 | 3 | 1 | 1 | 3 | 18 | 12 | 6 | 2 | 54
  Black or African American | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 5
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 3 | 3 | 1 | 4 | 20 | 12 | 6 | 2 | 60
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  centimeter (cm)
    number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 1 | 4 | 20 | 12 | 5 | 2 | 59
    (all) | 173.1 (9.63) | 167.5 (7.60) | 167.4 (4.54) | 180.1 (14.25) | 165.4 (7.90) | 178 (NA) — Standard deviation is not estimable for 1 participant. | 169.7 (12.18) | 165.8 (11.28) | 165.7 (13.26) | 169.3 (9.16) | 156.7 (6.08) | 167.5 (11.07)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 87.50 (12.560) | 71.03 (5.937) | 74.87 (5.036) | 109.90 (12.760) | 80.77 (2.542) | 82.3 (NA) — Standard deviation is not estimable for 1 participant. | 82.98 (21.532) | 77.81 (23.760) | 72.60 (15.579) | 93.20 (16.811) | 71.70 (36.770) | 80.27 (19.946)
Body Surface Area [Mean (Standard Deviation); unit: meter square] — Body Surface Area (m^2)=[Height(cm) * Weight (kg)]/3600)^1/2. Population: Here, number analyzed are the participants who were evaluated for this baseline measure.
  meter square
    number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 1 | 4 | 20 | 12 | 5 | 2 | 59
    (all) | 2.05 (0.192) | 1.82 (0.100) | 1.86 (0.062) | 2.34 (0.229) | 1.93 (0.071) | 2.02 (NA) — Standard deviation is not estimable for 1 participant. | 1.97 (0.335) | 1.88 (0.342) | 1.82 (0.237) | 2.09 (0.265) | 1.74 (0.495) | 1.92 (0.291)
Time Since Primary Diagnosis to First Dose [Median (Full Range); unit: months] | 59.1 [55 to 291] | 61.8 [57 to 94] | 45.8 [34 to 152] | 80.4 [46 to 88] | 38.4 [13 to 58] | 44.62 [44.62 to 44.62] | 35.2 [21 to 85] | 56.9 [19 to 124] | 42.7 [12 to 151] | 71.9 [61 to 97] | 76.1 [46 to 106] | 57.4 [12 to 291]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. An SAE is any untoward medical occurrence that results in death;is life-threatening;requires inpatient hospitalization or prolongation of present hospitalization;results in persistent or significant disability/incapacity;is a congenital anomaly/birth defect;or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent. A TEAE is defined as an AE that occurs after administration of first dose of study drug and through 30 days after last dose of study drug or until start of subsequent antineoplastic therapy.
Time Frame: From first dose of the study drug through 30 days after the last dose of study drug or start of subsequent antineoplastic therapy (Up to 81.1 months)
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Groups:
- Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2: Ixazomib 2.0 mg/m^2, capsule, orally, on Days 1, 4, 8 and 11 during a 21-day treatment cycle until progressive disease (PD) or unacceptable toxicity up to 12 months unless the investigator and sponsor determine the participant would benefit from therapy beyond 12 months. Participants with relapsed or refractory disease after >=1 prior therapy which must include thalidomide (or lenalidomide) and corticosteroid, but who never received a proteasome inhibitor.
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 20 | 12 | 6 | 2
Participants
  AEs | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 20 | 12 | 6 | 2
  SAEs | 0 | 0 | 2 | 2 | 0 | 5 | 3 | 14 | 6 | 3 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities Reported as TEAEs
Description: The number of participants with any clinically significant abnormal standard safety laboratory values collected throughout the study reported as TEAEs. Parameters assessed were hematology, serum chemistry and urinalysis.
Time Frame: as for outcome 1
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 20 | 12 | 6 | 2
Participants
  Blood Creatinine Increased | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0
  Blood Urea Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  White Blood Cell Count Decreased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Alanine Aminotransferase Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Liver Function Test Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood Calcium Increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Haematocrit Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Haemoglobin Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With a TEAE of Peripheral Neuropathy
Description: Neurotoxicity was assessed as the number of participants with the TEAE of peripheral neuropathy.
Time Frame: as for outcome 1
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 20 | 12 | 6 | 2
Participants
  Neuropathy Peripheral | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 0
  Peripheral Sensory Neuropathy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as TEAEs
Description: The number of participants with any clinically significant changes in vital signs collected throughout the study that were reported as TEAEs. Measurement of vital signs, included oral temperature, blood pressure, and heart rate.
Time Frame: as for outcome 1
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 7 | 4 | 20 | 12 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

5. Primary Outcome: Maximum Tolerated Dose (MTD) of Ixazomib
Description: MTD was highest dose of Ixazomib, at which <=1 of 6 participants experienced dose-limiting toxicity (DLT) during Cycle 1 of Phase 1. DLT was defined as any of following considered possibly related to therapy: Grade 4 neutropenia (absolute neutrophil count [ANC] <500 cell per cubic millimeter [cells/mm^3]) for >7 days;Grade 3 neutropenia with fever or infection; Grade 4 thrombocytopenia (platelets < 25,000/mm^3) for >7 days;Grade 3 thrombocytopenia with clinically significant bleeding; platelet count <10,000/mm^3; Grade 2 peripheral neuropathy with pain or >=Grade 3 peripheral neuropathy; >=Grade 3 nausea/emesis, diarrhea controlled by supportive therapy; Grade 3 QTc prolongation (QTc >500 millisecond [msec]);any >=Grade 3 nonhematologic toxicity except Grade 3 arthralgia/myalgia; or <1 week Grade 3 fatigue; delay in initiation of the subsequent therapy cycle by >2 weeks; other >=Grade 2 study drug-related nonhematologic toxicities requiring therapy discontinuation.
Time Frame: Cycle 1 (21 days)
Population: DLT-evaluable population was defined as all participants who received all Cycle 1 doses of ixazomib and completed Cycle 1 or who experienced DLT in Cycle 1.
Measure: Number; unit: mg/m^2
Groups:
- Ixazomib (All Groups): All participants who received ixazomib 0.24 mg/m^2, 0.48 mg/m^2, 0.8 mg/m^2, 1.2 mg/m^2, 1.68 mg/m^2, 2 mg/m^2 or 2.23 mg/m^2 in dose-escalation cohorts.
Arm/Group | Ixazomib (All Groups)
Number analyzed (Participants) | 26
mg/m^2 | 2

6. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Ixazomib
Description: The RP2D of Ixazomib was determined in Part 1 (dose escalation) on the basis of the totality of safety, tolerability, pharmacokinetics (PK) and pharmacodynamic data observed in Cycle 1 and beyond.
Time Frame: Cycle 1 through Cycle 39 (Up to 28.3 months)
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: mg/m^2
Arm/Group | Ixazomib (All Groups)
Number analyzed (Participants) | 26
mg/m^2 | 2

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (up to 264 hours) postdose
Population: PK population was defined as all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of ixazomib PK parameters. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 6 | 3 | 17 | 9 | 6 | 1
ng/mL
  Day 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 6 | 3 | 14 | 9 | 6 | 1
  Day 1 | 2.120 (0.3974) | 10.190 (2.5597) | 22.200 (11.3137) | 29.000 (24.1831) | 21.100 (10.1237) | 68.167 (34.7876) | 117.933 (67.1924) | 58.900 (36.1337) | 59.343 (41.9853) | 85.600 (58.8496) | 26.600 (NA) — SD was not calculated for 1 participant.
  Day 11: number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 5 | 2 | 14 | 7 | 5 | 1
  Day 11 | 2.837 (1.5051) | 8.857 (5.5598) | 31.650 (15.2028) | 56.500 (14.1421) | 101.100 (71.3597) | 85.420 (30.7632) | 105.450 (41.7900) | 59.871 (32.5851) | 61.800 (24.8780) | 109.660 (27.5668) | 27.200 (NA) — SD was not calculated for 1 participant.

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 264 hours) postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 6 | 3 | 17 | 9 | 6 | 1
hours
  Day 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 6 | 3 | 14 | 9 | 6 | 1
  Day 1 | 1.000 [0.57 to 2.00] | 1.000 [0.50 to 1.50] | 0.775 [0.55 to 1.00] | 0.775 [0.50 to 1.05] | 1.000 [1.00 to 2.02] | 1.000 [0.25 to 1.08] | 1.000 [0.72 to 1.08] | 1.000 [0.52 to 2.00] | 0.617 [0.50 to 3.97] | 0.525 [0.25 to 1.05] | 1.000 [1.00 to 1.00]
  Day 11: number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 5 | 2 | 14 | 7 | 5 | 1
  Day 11 | 1.100 [1.05 to 4.07] | 1.000 [0.50 to 1.17] | 1.275 [0.55 to 2.00] | 0.500 [0.50 to 0.50] | 1.000 [0.57 to 1.05] | 0.667 [0.50 to 1.50] | 0.832 [0.53 to 1.13] | 1.010 [0.50 to 23.60] | 0.583 [0.50 to 1.03] | 1.500 [0.62 to 1.53] | 1.500 [1.5 to 1.5]

9. Secondary Outcome: AUC(0-last): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 264 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 6 | 3 | 17 | 9 | 6 | 1
hr*ng/mL
  Day 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 3 | 6 | 2 | 12 | 9 | 5 | 1
  Day 1 | 3.383 (1.7210) | 20.700 (4.5255) | 109.000 (41.0122) | 159.050 (91.8532) | 251.000 (62.5060) | 449.000 (185.9516) | 416.500 (47.3762) | 418.175 (218.7115) | 351.000 (141.4337) | 410.000 (138.7732) | 509.000 (NA) — SD was not calculated for 1 participant.
  Day 11: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2 | 5 | 2 | 13 | 7 | 5 | 1
  Day 11 | 56.533 (15.5095) | 177.667 (115.6820) | 458.000 (42.4264) | 605.000 (NA) — SD was not calculated for 1 participant. | 808.500 (212.8391) | 1435.600 (1027.3881) | 1915.000 (148.4924) | 903.846 (382.9033) | 937.857 (334.2082) | 2297.200 (1137.8221) | 1010.000 (NA) — SD was not calculated for 1 participant.

10. Secondary Outcome: AUC(0-72): Area Under the Plasma Concentration-Time Curve From Time 0 to 72 Hours Postdose for Ixazomib
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 72 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 6 | 3 | 17 | 9 | 6 | 1
hr*ng/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 6 | 2 | 11 | 9 | 5 | 1
  Day 1 |  |  | 109.00 (41.012) | 159.05 (91.853) | 251.00 (62.506) | 449.00 (185.952) | 416.50 (47.376) | 451.64 (194.522) | 351.00 (141.434) | 410.00 (138.773) | 509.00 (NA) — SD was not calculated for 1 participant.
  Day 11: number analyzed (Participants) | 3 | 3 | 2 | 1 | 2 | 5 | 2 | 13 | 7 | 5 | 1
  Day 11 | 56.53 (15.509) | 177.67 (115.682) | 458.00 (42.426) | 605.00 (NA) — SD was not calculated for 1 participant. | 808.50 (212.839) | 1435.60 (1027.388) | 1915.00 (148.492) | 903.85 (382.903) | 937.86 (334.208) | 2297.20 (1137.822) | 1010.00 (NA) — SD was not calculated for 1 participant.

11. Secondary Outcome: λz: Terminal Disposition Phase Rate Constant for Ixazomib
Time Frame: Cycle 1, Day 11: predose and at multiple time points (Up to 264 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 0 | 1 | 0 | 2 | 3 | 5 | 2 | 11 | 7 | 4 | 1
1/hr |  | 0.005 (NA) — Standard deviation was not calculated for 1 participant. |  | 0.005 (0.0001) | 0.006 (0.0012) | 0.007 (0.0012) | 0.008 (0.0007) | 0.006 (0.0015) | 0.006 (0.0018) | 0.006 (0.0020) | 0.005 (NA) — Standard deviation was not calculated for 1 participant.

12. Secondary Outcome: T1/2: Terminal Disposition Phase Elimination Half-life for Ixazomib
Time Frame: Cycle 1, Day 11: predose and at multiple time points (up to 264 hours) postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 0 | 1 | 0 | 2 | 3 | 5 | 2 | 11 | 7 | 4 | 1
hr |  | 135.00 (NA) — Standard deviation was not calculated for 1 participant. |  | 126.50 (2.121) | 129.33 (25.658) | 105.88 (21.071) | 92.70 (8.485) | 115.85 (26.368) | 123.06 (33.877) | 124.93 (41.330) | 134.00 (NA) — Standard deviation was not calculated for 1 participant.

13. Secondary Outcome: CL/F: Blood Clearance Calculated Using the Observed Value of the Last Quantifiable Concentration for Ixazomib
Description: CL/F is apparent clearance of the drug from the plasma.
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 264 hours) postdose
Population: CL/F was not reported as this PK parameter could not be calculated.
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Emax: Maximum Observed Effect for Ixazomib
Description: Emax was determined to characterize the whole blood 20S proteasome inhibition parameters.
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 264 hours) postdose
Population: No data is reported due to concerns about the third-party laboratory's performance of the 20S assay that precluded the ability to confirm the accuracy of the data generated. The data was not considered reliable.
Groups:
- VELCADE-Relapsed Expansion Cohort: MLN9708 2.0 mg/m^2: Ixazomib (MLN9708) 2 mg/m^2 (MTD), capsule, orally, twice weekly on Days 1, 4, 8 and 11 in 21-day treatment cycles until PD or unacceptable toxicity in participants with relapsed multiple myeloma previously treated with VELCADE during Part 2 (dose expansion cohort) of the study.
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | VELCADE-Relapsed Expansion Cohort: MLN9708 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: TEmax: Time to Maximum Observed Effect (Emax) for Ixazomib
Description: TEmax was determined to characterize the whole blood 20S proteasome inhibition parameters.
Time Frame: Cycle 1, Days 1 and 11: Predose and at multiple time points (Up to 264 hours) postdose
Population: as for outcome 14
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with complete response (CR) or partial response (PR) or minimal response (MR) as assessed by the investigator using International Myeloma Working Group Uniform Response criteria. CR=Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow. PR=≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg /24 h. MR=25-49% reduction in the serum monoclonal paraprotein maintained for a minimum of 6 weeks; 50-89% reduction in 24-h urinary light chain excretion, which still exceeds 200 mg/24 h, maintained for a minimum of 6 weeks; for participants with non-secretory myeloma only, 25-49% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy, if biopsy is performed, maintained for a minimum of 6 weeks; 25-49% reduction in the size of soft tissue plasmacytomas; no increase in the size or number of lytic bone lesions.
Time Frame: Cycle 1 through Cycle 115 (Up to 80.1 months)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, had measurable disease at baseline, and at least 1 post baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 6 | 2 | 20 | 11 | 6 | 2
percentage of participants
  CR+PR | 0 | 0 | 0 | 33 | 0 | 0 | 50 | 5 | 9 | 33 | 0
  CR+PR+MR | 0 | 0 | 0 | 33 | 0 | 0 | 50 | 10 | 18 | 33 | 0

ADVERSE EVENTS:
Time Frame: From first dose of the study drug through 30 days after the last dose of study drug or start of subsequent antineoplastic therapy (Up to 81.1 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/3 | 0/7 | 0/4 | 1/20 | 0/12 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/3 | 2/3 | 0/3 | 5/7 | 3/4 | 14/20 | 6/12 | 3/6 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 7/7 | 4/4 | 20/20 | 12/12 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 (N=3) | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 (N=3) | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 (N=3) | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 (N=3) | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 (N=3) | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 (N=7) | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 (N=4) | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=20) | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=12) | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 (N=6) | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation Cohort 1: Ixazomib 0.24 mg/m^2 (N=3) | Dose Escalation Cohort 2: Ixazomib 0.48 mg/m^2 (N=3) | Dose Escalation Cohort 3: Ixazomib 0.8 mg/m^2 (N=3) | Dose Escalation Cohort 4: Ixazomib 1.2 mg/m^2 (N=3) | Dose Escalation Cohort 5: Ixazomib 1.68 mg/m^2 (N=3) | Dose Escalation Cohort 6: Ixazomib 2.0 mg/m^2 (N=7) | Dose Escalation Cohort 7: Ixazomib 2.23 mg/m^2 (N=4) | Relapsed and Refractory Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=20) | Velcade-Relapsed (VR) Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=12) | Proteasome Inhibitor-Naive Expansion Cohort: Ixazomib 2 mg/m^2 (N=6) | Carfilzomib Expansion Cohort: Ixazomib 2.0 mg/m^2 (N=2)
Fatigue (General disorders) | 1 | 2 | 1 | 1 | 2 | 4 | 2 | 12 | 8 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 4 | 2 | 3 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 8 | 3 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 4 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 4 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 1 | 1 | 4 | 1 | 6 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 3 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 6 | 7 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cranial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5 | 3 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 6 | 5 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 3 | 7 | 8 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 3 | 3 | 4 | 6 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 4 | 5 | 4 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 3 | 9 | 3 | 3 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.